CLINICAL TRIAL: NCT01659528
Title: Establishing Nomograms of Penile Length and Width Throughout the Weeks of Pregnancy - A Prospective Descriptive Study.
Brief Title: Establishing Nomograms of Penile Length and Width Throughout the Weeks of Pregnancy
Status: Withdrawn | Type: Observational
Why Stopped: A similar article was already published by another investigator.
Sponsor: Carmel Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: CMC-11-0028-CTIL
Record Dates: First submitted 2012-08-05; First posted 2012-08-07 (Estimated); Last update posted 2013-02-01 (Estimated); Status verified 2013-01

CONDITIONS: Micropenis
Keywords: Penis; Micropenis; Nomograms; Ultrasound; Fetus
MeSH Terms: conditions — Penis agenesis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to establish nomograms of penile length and width throughout the weeks of pregnancy.

DETAILED DESCRIPTION:
Identifying pathology of male genitalia is important. It can be an isolated pathology, or connected to disorders in other organs, as part of genetic syndromes or endocrine disorders. Micropenis is a disorder, which is important to diagnose in the womb. Micropenis is defined as a penis which is measured 2.5 standard deviation below average. It is also thinner by diameter. This finding can also be the first expression of a lethal hormonal deficiency, hence the reason for early detection by ultrasound during pregnancy.

Past prenatal diagnosis ultrasound studies, measured the penis from the scrotum to the tip of the penis. Another study evaluated formalin fixated fetuses after pregnancy terminations, in which the penis was measured from the abdominal wall to the tip of the penis. To date there are no nomograms for penile length, via ultrasound measurement from abdominal wall or for penile width. The investigators assume that measuring the penis from the abdominal wall is more accurate and standard than from the end of the scrotum, which is a less definitive reference point.

The investigators aim to establish nomograms of penile length throughout the weeks of pregnancy. Exceptional penile width can also point out a problem with male genitalia. Therefore the investigators wish, as well to establish nomograms of penile width.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy
* Proper pregnancy dating
* Normal fetal anatomical scan
* Gestational age 14 to 37 weeks
* Women aged 18 to 50

Exclusion Criteria:

* Multiple pregnancy
* Gestational age under 14 or above 37 weeks
* Fetus Small or Large for gestational age
* Abnormal anatomical scan or women who didn't perform such scan
* Minors

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant women addressing for routine ultrasound scan at the ultrasound unit.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2012-07; Primary Completion 2014-07 (Estimated); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
Penile length | between 14 and 37 weeks gestation
Penile width | between 14 and 37 weeks gestation

CONTACTS AND LOCATIONS:
Overall Officials: Yael Goldberg, MD, Principal Investigator — Head of Obstetrics and Gynecologic Ultrasound Unit, The Lady Davis Carmel Medical Center, Affiliated with the Rappaport Faculty of Medicine, Technion, Haifa, Israel
Locations (1):
- OBGYN Ultrasound Unit, Carmel Medical Center, Haifa, Israel, Israel

REFERENCES:
- [Background] Achiron R, Pinhas-Hamiel O, Zalel Y, Rotstein Z, Lipitz S. Development of fetal male gender: prenatal sonographic measurement of the scrotum and evaluation of testicular descent. Ultrasound Obstet Gynecol. 1998 Apr;11(4):242-5. doi: 10.1046/j.1469-0705.1998.11040242.x. PMID 9618845
- [Background] Feldman KW, Smith DW. Fetal phallic growth and penile standards for newborn male infants. J Pediatr. 1975 Mar;86(3):395-8. doi: 10.1016/s0022-3476(75)80969-3. PMID 1113226
- [Background] Aaronson IA. Micropenis: medical and surgical implications. J Urol. 1994 Jul;152(1):4-14. doi: 10.1016/s0022-5347(17)32804-5. No abstract available. PMID 8201683
- [Background] Toppari J, Kaleva M, Virtanen HE. Trends in the incidence of cryptorchidism and hypospadias, and methodological limitations of registry-based data. Hum Reprod Update. 2001 May-Jun;7(3):282-6. doi: 10.1093/humupd/7.3.282. PMID 11392374